CLINICAL TRIAL: NCT04715945
Title: Southampton Women's Survey - a Study of Non-pregnant Women and Follow-up of Offspring Through Pregnancy and Childhood
Brief Title: Southampton Women's Survey
Acronym: SWS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: 276/97
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Child Development; Child Obesity; Child Behavior; Nutritional and Metabolic Diseases; Asthma in Children; Cardiovascular Risk Factor; Bone Loss
MeSH Terms: conditions — Pediatric Obesity; Child Behavior; Nutritional and Metabolic Diseases; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, mouth swaps, umbilical cord, cord blood, placental samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women: 12,583 women recruited when non-pregnant
- Children: 3,158 liveborn singleton offspring of women recruited to the study

SUMMARY:
The Southampton Women's Survey was established to assess the influence of factors operating before conception and during pregnancy on the health and development of the offspring. 12,583 non-pregnant young women were recruited, and 3,158 were followed through pregnancy, with their offspring followed-up at 6 months and 1, 2, 3, 4, 6-7, 8-9 and 12-13 years. The 17-19 year follow-up has been piloted and is about to start.

DETAILED DESCRIPTION:
The Southampton Women's Survey (SWS) was established to assess the influence of factors operating before conception and during pregnancy on the health and development of the offspring. 12,583 non-pregnant young women were recruited and the subsequent offspring of 3158 of them are being followed-up. Few other longitudinal studies of children have data on the tempo of prenatal growth, and none in high-income countries has information recorded before pregnancy.

The objectives of the SWS are: (a) to characterise the influences of a mother's own fetal growth and of her dietary balance, body composition and endocrine profile before and during pregnancy on (i) the early trajectory of fetal growth; (ii) the maintenance of this growth trajectory in late gestation; and (iii) placental and fetal adaptive responses, (b) to examine how maternal and intrauterine influences interact with the offspring's genes and postnatal environment to determine: (i) weight gain and linear catch-up growth in infancy; (ii) the pathways of growth and development during childhood that lead to poor adult health (obesity, obstructive airways disease, cardiovascular disease, diabetes, and osteoporosis).

Between 1998 and 2002, 12,583 women aged 20 to 34 years were interviewed and their diet, body composition, physical activity levels, lifestyles and social circumstances were assessed. Blood, urine and mouthwash samples were collected for genetic and other analyses. Women who subsequently became pregnant were followed-up at 11, 19 and 34 weeks' gestation and fetal ultrasound scans were performed to obtain longitudinal measurements of fetal growth during pregnancy. Between 1998 and 2007, 3,158 women delivered a single live born infant. Biological samples were taken and anthropometric measurements of the baby were made within 48 hours of birth. In a sample of 1,000 children, dual-energy X-ray absorptiometry (DXA) was performed in the first two weeks of life.

The children were followed up at ages 6, 12, 24 and 36 months. A variety of assessments were made at the different follow-up interviews including breastfeeding, diet, anthropometry, and illnesses. At 24 months, the social circumstances of the family were assessed and, at 36 months, parenting, and emotional and behavioural issues were recorded. Subsequently, samples of the cohort have been seen at specific ages; at 4 years approximately 1,000 cohort participants; at 6-7 years approximately 2,000, and at 8-9 years approximately 1,000. At each time point from 4 years, body composition and bone indices were assessed using DXA; at 4 years, cognitive function was measured, at 6-7 years the focus was respiratory health and cognitive function, and at 8-9 years cardiovascular structure and function. Over 1000 child have been seen at age 12-13 years and the visits at 17-19 years of age have been piloted and are about to start with a focus on preparation for parenthood. Furthermore, plans are being developed to follow up the 12,583 women originally recruited to the SWS to assess the influence of their younger adult lifestyles, body composition and hormones on their transition through the menopause.

ELIGIBILITY:
Inclusion Criteria:

* Not pregnant, resident in Southampton UK.

Exclusion Criteria:

* GP requested no contact

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Non-pregnant women
Study Population: All non-pregnant women in the correct age group living in Southampton between 1998 and 2002 were eligible.
Sampling Method: Non-Probability Sample
Enrollment: 12583 (Actual)
Dates: Start 1998-04-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Child health and development | 0 - 19 years
  Child health and development from birth to 19 years, focussing on body composition, nutrition, asthma and cardiovascular health

CONTACTS AND LOCATIONS:
Overall Officials: Cyrus Cooper, FMedSci, Study Director — University of Southampton

IPD SHARING:
Plan to Share IPD: Yes
All data can be shared subject to approval of SWS oversight group and completion of confidentiality agreements.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Most data are already available and will continue to be available we hope beyond completion of the study.
Access Criteria: Application to SWS oversight group
URL: http://www.mrc.soton.ac.uk/sws/

REFERENCES:
- [Result] Inskip HM, Godfrey KM, Robinson SM, Law CM, Barker DJ, Cooper C; SWS Study Group. Cohort profile: The Southampton Women's Survey. Int J Epidemiol. 2006 Feb;35(1):42-8. doi: 10.1093/ije/dyi202. Epub 2005 Sep 29. No abstract available. PMID 16195252
- [Derived] El-Heis S, Crozier SR, Loo EX, Tham EH, Harvey NC, Inskip HM; Southampton Women's Survey Study Group; Godfrey KM. Maternal Dietary Inflammatory Status and Serum Neopterin During Pregnancy: Influence on Infantile Atopic Eczema in the Offspring. Clin Transl Allergy. 2025 Jul;15(7):e70080. doi: 10.1002/clt2.70080. PMID 40714954
- [Derived] Simpson RF, Hesketh KR, Crozier SR, Baird J, Cooper C, Godfrey KM, Harvey NC, Westgate K, Inskip HM, van Sluijs EMF. The association between number and ages of children and the physical activity of mothers: Cross-sectional analyses from the Southampton Women's Survey. PLoS One. 2022 Nov 16;17(11):e0276964. doi: 10.1371/journal.pone.0276964. eCollection 2022. PMID 36383511